CLINICAL TRIAL: NCT05568953
Title: An Experimental Medicine Decipher of a Minimum Correlate of Cellular Immunity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: JEYF-Tcell-001
Record Dates: First submitted 2022-08-29; First posted 2022-10-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Infectious Disease; Yellow Fever; Japanese Encephalitis; Viral Infection
Keywords: Yellow Fever; Japanese Encephalitis; YF17D; JE-YF17D; T-cell Immunity; Cellular Immunity; Live-attenuated Vaccines
MeSH Terms: conditions — Communicable Diseases; Yellow Fever; Encephalitis, Japanese; Virus Diseases

STUDY DESIGN:
Intervention Model Description: 58 subjects will be randomised into 1 of 2 arms (Arm B1 and Arm B2) in a 1:1 ratio, in a double-blind fashion. Randomization will be performed via a web-based randomization system: http://www.randomization.com by an independent person who has no direct contact with the subjects. Randomization opaque envelopes will be prepared by an independent team in accordance to the Master Randomization List generated. The randomization envelopes are to be opened sequentially for each enrollment by the study team and will determine the subject's allocation to one of the three groups.
  Arm B3 will be conducted as a separate single-arm open label design in 14 subjects.
  Enrolled subjects will be randomised into 1 of 3 arms (Arm B1, Arm B2 and Arm B3) in a 2:2:1 ratio. The study will be double-blinded.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Arms B1 and B2 will be double-blinded. Arm B3 will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (JE-YF17D vaccine followed by YF17D vaccine) (Experimental): 28 subjects will receive one dose of the JE-YF17D vaccine (Imojev, Sanofi Pasteur, 0.5mls (4.0 - 5.8 log plaque forming units [PFU])) on Day 0 followed by one dose of the YF17D vaccine (Stamaril, Sanofi Pasteur, 0.5mls (3 - 4 log PFU) ) on Day 28.
  Interventions: Biological: Stamaril; Biological: Imojev
- Arm 2 (YF17D vaccine followed by JE-YF17D vaccine) (Experimental): 28 subjects will receive one dose of the YF17D vaccine (Stamaril, Sanofi Pasteur, 0.5mls (3 - 4 log PFU)) on Day 0 followed by one dose of the JE-YF17D vaccine (Imojev, Sanofi Pasteur, 0.5mls (4.0 - 5.8 log plaque forming units [PFU]) on Day 28.
  Interventions: Biological: Stamaril; Biological: Imojev
- Arm 3 (Inactivated JE vaccine followed by YF17D vaccine) (Experimental): 14 subjects will receive one dose of the inactivated JE vaccine (Ixiaro, Valneva, 0.5mls) on Day 0 followed by one dose of the YF17D vaccine (Stamaril, Sanofi Pasteur, 0.5mls (3 - 4 log PFU)) on Day 28.
  Interventions: Biological: Stamaril; Biological: Ixiaro

INTERVENTIONS:
Biological: Stamaril — Stamaril is licensed by the Health Sciences Authority (HSA), Singapore. The vaccine are manufactured by Sanofi Pasteur and sourced from Sanofi Pasteur's local distributor.
  Other Names: YF17D vaccine
Biological: Imojev — Imojev is licensed by the Health Sciences Authority (HSA), Singapore. The vaccine are manufactured by Sanofi Pasteur and sourced from Sanofi Pasteur's local distributor.
  Other Names: JE-YF17D vaccine
  Arms: Arm 1 (JE-YF17D vaccine followed by YF17D vaccine); Arm 2 (YF17D vaccine followed by JE-YF17D vaccine)
Biological: Ixiaro — Ixiaro is licensed by the Health Sciences Authority (HSA), Singapore. The Ixiaro vaccines are manufactured by Valneva and sourced from local distributor, Aenon Pharmaceuticals SEA Pte Ltd.
  Other Names: Inactivated Japanese Encephalitis vaccine
  Arms: Arm 3 (Inactivated JE vaccine followed by YF17D vaccine)

SUMMARY:
We hypothesize that a high CD4+ and CD8+ T cell count will reduce viremia upon challenge with a structurally heterologous virus, and correspondingly result in reduced magnitude of host response to challenge infection.

Primary Objective: To compare, after challenge with a structurally heterologous vaccine, the differences in levels of viremia between healthy adults who received primary vaccination with either YF17D vaccine, chimeric JE-YF17D vaccine, or inactivated JE vaccine.

58 subjects will be randomised into 1 of 2 arms (Arm B1 and Arm B2) in a 1:1 ratio, in a double-blind fashion. Subjects in Arm B1 will receive JE-YF17D vaccine (Imojev, Sanofi Pasteur) on Day 0 followed by YF17D vaccine (Stamaril, Sanofi Pasteur) on Day 28. Subjects in Arm B2 will receive Stamaril on Day 0 followed by Imojev on Day 28. Arm B3 will be conducted as a separate single-arm open label design in 14 subjects. Subjects in Arm B3 will receive inactivated JE vaccine (Ixiaro, Valneva) on Day 0 followed by Stamaril on Day 28.

The rationale for these three study arms is as follows: Arm B1 will show the impact low levels of viremia, and the resultant low levels of virus-specific CD4+ and CD8+ T cells, would have on YF17D infection. In contrast, YF17D vaccination in Arm B2 would produce high levels of viremia, and in turn high levels virus-specific T cells, thus likely ameliorating JE-YF17D infection. Arm B3 will serve as the control arm, as vaccination with inactivated JE vaccine would not produce any YF17D-specific T cell response. Notably, the first vaccination in Arms B1 and B2 would also provide the viremia response in the absence of virus-specific T cells, which would serve as a reference point to interpret the outcome of the second vaccination.

DETAILED DESCRIPTION:
Criteria for Recruitment and Recruitment Process: Subjects will be recruited from SingHealth Investigational Medicine Unit (IMU) healthy volunteer database and recruitment posters. Subjects will be given a copy of the Participant Information and Informed Consent Form to read upon their arrival. A briefing session on the study will be conducted by the Investigator. Thereafter, subjects will be ushered into a private room where informed consent is obtained and where questions about the study can be asked freely. Subjects will not be rushed into making a decision to participate in the study. They will be encouraged to speak to their family members about participation in the study; and allowed to defer their decision (without any prejudice) to participate till after discussion with their family members.

Screening Visits and Procedures: Subjects will be recruited via the SingHealth Investigational Medicine Unit (IMU). Informed written consent will be sought from subjects who fulfill criteria for enrollment. All consented subjects will undergo screening, which includes physical examination, full blood count, liver function test, anti-dengue antibodies ELISA (Enzyme-Linked Immunosorbent Assay) and urinary pregnancy test (for female subjects of child-bearing potential).

A urine pregnancy test will be performed at screening and on the day of vaccination (day 0 and day 28) for female subjects of child-bearing potential. Only those with a negative urine pregnancy test will be considered to be eligible for the study, provided that other eligibility criteria were fulfilled.

Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) must agree to use adequate and reliable contraceptive measures (e.g. spermicides, condoms, contraceptive pills) or practice abstinence for 10 days after vaccination.

Study Visits and Procedures: 58 subjects will be randomised into 1 of 2 arms (Arm B1 and Arm B2) in a 1:1 ratio, in a double-blind fashion. Subjects in Arm B1 will receive JE-YF17D vaccine (Imojev, Sanofi Pasteur) on Day 0 followed by YF17D vaccine (Stamaril, Sanofi Pasteur) on Day 28. Subjects in Arm B2 will receive Stamaril on Day 0 followed by Imojev on Day 28. Arm B3 will be conducted as a separate single-arm open label design in 14 subjects. Subjects in Arm B3 will receive inactivated JE vaccine (Ixiaro, Valneva) on Day 0 followed by Stamaril on Day 28. Study visits in all arms will occur on Day 0, 4, 7, 10, 14, 28, 29, 32, 35, 38, 42, 58. At each study visit, physical examination, vital signs and research blood sampling will be performed. On Day 0 and Day 28, blood sampling will be performed prior to vaccination.

Final study visit: Last study visit will be on Day 58 post-study vaccination.

Post study follow up and procedures: There is no requirement for post-study follow-up or procedures.

Safety Monitoring Plan: The study may be evaluated by government inspectors/ regulatory authorities who must be allowed access to e-CRFs, source documents, and other study files. The inspectors will review CRFs and compare them with source documents to verify accurate and complete collection of data and confirm that the study is being conducted according to the protocol, ICH Good Clinical Practices (ICH-GCP) and all applicable regulations.

At any time post-vaccination, all subjects will be trained to observe for systemic AEs. A diary will also be given to the subjects to record such events should they occur during this period. Should they develop systemic symptoms that require intervention, they will report to the study site for medical evaluation and receive the appropriate therapy. Duration of symptoms will be recorded. Any concomitant medication use during this period will also be recorded.

During the study, full history taking and physical examination will be performed at both scheduled and unscheduled visits. A full physical examination will only be done at the screening visit, while a brief physical examination will be done for all subsequent visits. The Common Terminology Criteria for Adverse Events (CTCAE), routinely employed in clinical trials, will be used to define AE terminology and severity. Management of AEs is at the discretion of the study team PI and co-Is, guided by severity and clinical indication for intervention. All medication prescribed for the management of AEs will be documented in the medication/concomitant medication clinical record form. Details of AE event terminology, date and time of event start and end, severity, using the CTCAE or treatment given, impact on work and to the continuation of the study, and final outcome of the event will be recorded on the case report until resolution of the event.

Data Quality Assurance: The PI and Co-Is will review the study periodically for data and safety monitoring. Internal quality checks will be performed by two CRCs who are study team members. The data entered by one CRC will be checked by another using the source documents. The study may also be picked for monitoring by SingHealth Office of Research Integrity and Compliance (ORIC) or evaluated by government inspectors/regulatory authorities who must be allowed access to e-CRFs, source documents, and other study files. The monitors/inspectors may review CRFs and compare them with source documents to verify accurate and complete collection of data and confirm that the study is being conducted according to the protocol, ICH-Good Clinical Practices (ICH-GCP) and all applicable regulations.

Data Entry and Storage: All participant's data will be de-identified upon recruitment. Hardcopy research data collection forms such as CRFs, logs and diaries will be kept in the Investigator's Site File and stored in SingHealth IMU under lock and key, accessible only to delegated study team members.

Direct data capture of demographic and clinical data will be captured on source documents. Identifiers will be kept in a separate file in another office and every effort will be made to protect the privacy of the participants. The data to be analysed will contain only de-identified data. An electronic data capture system will be used. All electronic data will be password protected and can only be accessed by study team members. Specimens, test results or pathogen data will be stored at Duke-NUS EID laboratory in a stand-alone PC whereby access is password protected.

Determination of sample size: To detect an effect size of 0.8 SD in mean viremia level on log(10) scale between first and second with the same vaccine - first dose of will be analysed against those who received YF17D after JE-YF17D and vice versa - a sample size of 25 per group will provide 80% power at 5% two-sided type 1 error rate. To allow for 10% early dropouts, a total sample size of 28 per group for Arm B1 and B2 is targeted. For Arm B3, which is the control group, a sample size of 14 will be used.

Statistical and Analytical plan: Distributional diagnostic plots will be used to examine the shape of distributions of T-cell counts immediately before the challenge vaccination and the subsequent vaccine viremia. Parametric (t-test) or non-parametric (Mann-Whitney U) procedures will be used to assess the differences in T-cell counts and the various measured variables such as viremia, antibody titres and cytokine levels. Pearson's or Spearman's correlation coefficients will be used, as appropriate, to examine the association between T-cell levels and these variables.

The frequency of symptoms reported and the type of symptoms will first be analysed by determining the median and the interquartile ranges. We will then analyse how the first vaccination impact the symptomatic outcome of the challenge vaccination using 2x2 tables and chi square analysis or Fisher's exact test, whichever is appropriate. Parametric (t-test) or non-parametric (Mann-Whitney U) procedures will be used to assess the differences in pre-challenge virus-specific T-cell counts among those with symptoms and those without.

Tests which will be performed on the blood samples: DENV IgG ELISA, FBC, Liver Panel, Viremia (NS5 PCR), cytokines, Anti-NS1 Ab, T-cell studies (AIM, ELLISPOT, ELLA), BCR sequencing, PRNT and gene expression.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults, 21-45 years of age at time of screening
2. Willing to comply to study procedures and adhere to study schedule visits.
3. Satisfactory baseline medical assessment as assessed by physical examination and a stable health status. The laboratory values must be within the normal range of the assessing site or show abnormalities that are deemed not clinically significant as judged by the investigator. A stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event.
4. Accessible vein for blood collection.
5. Ability to provide informed consent.
6. Female subjects of non-child bearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Post-menopausal subjects must have had at least 12 months of natural (spontaneous) amenorrhea
7. Female subjects of child bearing potential with negative urine pregnancy tests on the day of screening and vaccination.
8. Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) must agree to use adequate and reliable contraceptive measures (e.g. spermicides, condoms, contraceptive pills) or practice abstinence for 10 days after vaccination.

Exclusion Criteria:

1. History of presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, haematological, endocrine or immunosuppressive disorders that would be a risk factor when administered the investigational product (IP)
2. Previous receipt of Imojev, Stamaril or Ixiaro vaccines, or any other yellow fever or Japanese encephalitis vaccines
3. Previous history of Yellow fever virus or Japanese encephalitis infection
4. Known allergy to Imojev, Stamaril or Ixiaro vaccines or their components
5. History of severe food/drug/vaccine allergies e.g. angioedema, anaphylaxis
6. Known allergy to egg or egg products
7. History of thymus gland disease
8. Diagnosed with cancer or on treatment for cancer (with the exception of localized basal cell carcinoma) within 3 years prior to screening
9. Evidence of clinically significant anemia (Hb <10 g/dl)
10. Blood donation exceeding >450mls in the past 3 months
11. Presence of acute infection in the preceding 7 days or presence of a temperature ≥ 38.0°C (oral or tympanic temperature assessment), or acute symptoms greater than of "mild" severity on the scheduled date of first dose
12. Woman who is pregnant or breast feeding
13. Evidence of substance abuse, or previous substance abuse including alcohol
14. Participation in a study involving administration of an investigational compound (including investigational vaccines) within the past three months, or planned participation during the duration of this study.
15. Receipt of anti-inflammatory drugs (such as NSAIDs or systemic steroids) in the past 7 days.
16. Receipt of any licensed vaccine in the past 30 days before the first study vaccine dose.
17. Positive serum Dengue IgG by ELISA
18. Any condition that, in the opinion of the investigator, would complicate or compromise the study or wellbeing of the subject.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Viremia levels after second vaccination | Day 0 to Day 58
  Viremia level (genome copies/ml) after second vaccination with either JE-YF17D or YF17D

SECONDARY OUTCOMES:
T cell responses after vaccination | Day 0 to Day 58
  Magnitude of antigen-specific T cell responses after vaccination.
Viremia level after first vaccination | Day 0 to Day 58
  Viremia level after first vaccination with either JE-YF17D or YF17D
Duration of viremia after second vaccination | Day 0 to Day 58
  Duration (in days) of detectable viremia after second vaccination with either JEYF17D or YF17D.
Antibody Titres | Day 0 to Day 58
  Neutralising Antibody titres as measured by plaque reduction neutralisation test (PRNT50 and PRNT90) i.e the serum titer required to reduce viral plaques by 50% or 90% respectively, after second vaccination with either YF17D, JEYF17D or inactivated JE-YF17D vaccines.
Rates of Adverse Events | Day 0 to Day 58
  Rates of adverse events after vaccination with either JE-YF17D or YF17D

OTHER OUTCOMES:
Innate Immune Gene Expression | Day 0 to Day 58
  Levels of innate immune gene expression after vaccination with JE-YF17D, YF17D or inactivated JE vaccine.
Cytokine levels | Day 0 to 58
  Levels of cytokines after vaccination with JE-YF17D, YF17D or inactivated JE vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Kalimuddin, MRCP (UK), Principal Investigator — Singapore General Hospital
Locations (1):
- SingHealth Investigational Medicine Unit, Singapore, Singapore

REFERENCES:
- [Background] Braciale TJ, Hahn YS. Immunity to viruses. Immunol Rev. 2013 Sep;255(1):5-12. doi: 10.1111/imr.12109. PMID 23947343
- [Background] Smith CM, Wilson NS, Waithman J, Villadangos JA, Carbone FR, Heath WR, Belz GT. Cognate CD4(+) T cell licensing of dendritic cells in CD8(+) T cell immunity. Nat Immunol. 2004 Nov;5(11):1143-8. doi: 10.1038/ni1129. Epub 2004 Oct 10. PMID 15475958
- [Background] Luckheeram RV, Zhou R, Verma AD, Xia B. CD4(+)T cells: differentiation and functions. Clin Dev Immunol. 2012;2012:925135. doi: 10.1155/2012/925135. Epub 2012 Mar 14. PMID 22474485
- [Background] Valbon SF, Condotta SA, Richer MJ. Regulation of effector and memory CD8(+) T cell function by inflammatory cytokines. Cytokine. 2016 Jun;82:16-23. doi: 10.1016/j.cyto.2015.11.013. Epub 2015 Dec 10. PMID 26688544
- [Background] Oja AE, Saris A, Ghandour CA, Kragten NAM, Hogema BM, Nossent EJ, Heunks LMA, Cuvalay S, Slot E, Linty F, Swaneveld FH, Vrielink H, Vidarsson G, Rispens T, van der Schoot E, van Lier RAW, Ten Brinke A, Hombrink P. Divergent SARS-CoV-2-specific T- and B-cell responses in severe but not mild COVID-19 patients. Eur J Immunol. 2020 Dec;50(12):1998-2012. doi: 10.1002/eji.202048908. Epub 2020 Nov 16. PMID 33073359
- [Background] Sekine T, Perez-Potti A, Rivera-Ballesteros O, Stralin K, Gorin JB, Olsson A, Llewellyn-Lacey S, Kamal H, Bogdanovic G, Muschiol S, Wullimann DJ, Kammann T, Emgard J, Parrot T, Folkesson E; Karolinska COVID-19 Study Group; Rooyackers O, Eriksson LI, Henter JI, Sonnerborg A, Allander T, Albert J, Nielsen M, Klingstrom J, Gredmark-Russ S, Bjorkstrom NK, Sandberg JK, Price DA, Ljunggren HG, Aleman S, Buggert M. Robust T Cell Immunity in Convalescent Individuals with Asymptomatic or Mild COVID-19. Cell. 2020 Oct 1;183(1):158-168.e14. doi: 10.1016/j.cell.2020.08.017. Epub 2020 Aug 14. PMID 32979941
- [Background] Gallais F, Velay A, Nazon C, Wendling MJ, Partisani M, Sibilia J, Candon S, Fafi-Kremer S. Intrafamilial Exposure to SARS-CoV-2 Associated with Cellular Immune Response without Seroconversion, France. Emerg Infect Dis. 2021 Jan;27(1):113-21. doi: 10.3201/eid2701.203611. Epub 2020 Dec 1. PMID 33261718
- [Background] Seow J, Graham C, Merrick B, Acors S, Pickering S, Steel KJA, Hemmings O, O'Byrne A, Kouphou N, Galao RP, Betancor G, Wilson HD, Signell AW, Winstone H, Kerridge C, Huettner I, Jimenez-Guardeno JM, Lista MJ, Temperton N, Snell LB, Bisnauthsing K, Moore A, Green A, Martinez L, Stokes B, Honey J, Izquierdo-Barras A, Arbane G, Patel A, Tan MKI, O'Connell L, O'Hara G, MacMahon E, Douthwaite S, Nebbia G, Batra R, Martinez-Nunez R, Shankar-Hari M, Edgeworth JD, Neil SJD, Malim MH, Doores KJ. Longitudinal observation and decline of neutralizing antibody responses in the three months following SARS-CoV-2 infection in humans. Nat Microbiol. 2020 Dec;5(12):1598-1607. doi: 10.1038/s41564-020-00813-8. Epub 2020 Oct 26. PMID 33106674
- [Background] Long QX, Tang XJ, Shi QL, Li Q, Deng HJ, Yuan J, Hu JL, Xu W, Zhang Y, Lv FJ, Su K, Zhang F, Gong J, Wu B, Liu XM, Li JJ, Qiu JF, Chen J, Huang AL. Clinical and immunological assessment of asymptomatic SARS-CoV-2 infections. Nat Med. 2020 Aug;26(8):1200-1204. doi: 10.1038/s41591-020-0965-6. Epub 2020 Jun 18. PMID 32555424
- [Background] Ibarrondo FJ, Fulcher JA, Goodman-Meza D, Elliott J, Hofmann C, Hausner MA, Ferbas KG, Tobin NH, Aldrovandi GM, Yang OO. Rapid Decay of Anti-SARS-CoV-2 Antibodies in Persons with Mild Covid-19. N Engl J Med. 2020 Sep 10;383(11):1085-1087. doi: 10.1056/NEJMc2025179. Epub 2020 Jul 21. No abstract available. PMID 32706954
- [Background] Channappanavar R, Fett C, Zhao J, Meyerholz DK, Perlman S. Virus-specific memory CD8 T cells provide substantial protection from lethal severe acute respiratory syndrome coronavirus infection. J Virol. 2014 Oct;88(19):11034-44. doi: 10.1128/JVI.01505-14. Epub 2014 Jul 23. PMID 25056892
- [Background] Zhao J, Alshukairi AN, Baharoon SA, Ahmed WA, Bokhari AA, Nehdi AM, Layqah LA, Alghamdi MG, Al Gethamy MM, Dada AM, Khalid I, Boujelal M, Al Johani SM, Vogel L, Subbarao K, Mangalam A, Wu C, Ten Eyck P, Perlman S, Zhao J. Recovery from the Middle East respiratory syndrome is associated with antibody and T-cell responses. Sci Immunol. 2017 Aug 4;2(14):eaan5393. doi: 10.1126/sciimmunol.aan5393. Epub 2017 Aug 4. PMID 28778905
- [Background] Le Bert N, Tan AT, Kunasegaran K, Tham CYL, Hafezi M, Chia A, Chng MHY, Lin M, Tan N, Linster M, Chia WN, Chen MI, Wang LF, Ooi EE, Kalimuddin S, Tambyah PA, Low JG, Tan YJ, Bertoletti A. SARS-CoV-2-specific T cell immunity in cases of COVID-19 and SARS, and uninfected controls. Nature. 2020 Aug;584(7821):457-462. doi: 10.1038/s41586-020-2550-z. Epub 2020 Jul 15. PMID 32668444
- [Background] Yauch LE, Zellweger RM, Kotturi MF, Qutubuddin A, Sidney J, Peters B, Prestwood TR, Sette A, Shresta S. A protective role for dengue virus-specific CD8+ T cells. J Immunol. 2009 Apr 15;182(8):4865-73. doi: 10.4049/jimmunol.0801974. PMID 19342665
- [Background] Prestwood TR, Morar MM, Zellweger RM, Miller R, May MM, Yauch LE, Lada SM, Shresta S. Gamma interferon (IFN-gamma) receptor restricts systemic dengue virus replication and prevents paralysis in IFN-alpha/beta receptor-deficient mice. J Virol. 2012 Dec;86(23):12561-70. doi: 10.1128/JVI.06743-11. Epub 2012 Sep 12. PMID 22973027
- [Background] Bassi MR, Kongsgaard M, Steffensen MA, Fenger C, Rasmussen M, Skjodt K, Finsen B, Stryhn A, Buus S, Christensen JP, Thomsen AR. CD8+ T cells complement antibodies in protecting against yellow fever virus. J Immunol. 2015 Feb 1;194(3):1141-53. doi: 10.4049/jimmunol.1402605. Epub 2014 Dec 24. PMID 25539816
- [Background] Shrestha B, Pinto AK, Green S, Bosch I, Diamond MS. CD8+ T cells use TRAIL to restrict West Nile virus pathogenesis by controlling infection in neurons. J Virol. 2012 Sep;86(17):8937-48. doi: 10.1128/JVI.00673-12. Epub 2012 Jun 27. PMID 22740407
- [Background] Shrestha B, Diamond MS. Fas ligand interactions contribute to CD8+ T-cell-mediated control of West Nile virus infection in the central nervous system. J Virol. 2007 Nov;81(21):11749-57. doi: 10.1128/JVI.01136-07. Epub 2007 Sep 5. PMID 17804505
- [Background] Jain N, Oswal N, Chawla AS, Agrawal T, Biswas M, Vrati S, Rath S, George A, Bal V, Medigeshi GR. CD8 T cells protect adult naive mice from JEV-induced morbidity via lytic function. PLoS Negl Trop Dis. 2017 Feb 2;11(2):e0005329. doi: 10.1371/journal.pntd.0005329. eCollection 2017 Feb. PMID 28151989
- [Background] Shrestha B, Ng T, Chu HJ, Noll M, Diamond MS. The relative contribution of antibody and CD8+ T cells to vaccine immunity against West Nile encephalitis virus. Vaccine. 2008 Apr 7;26(16):2020-33. doi: 10.1016/j.vaccine.2008.02.009. Epub 2008 Feb 20. PMID 18339459
- [Background] Moodie Z, Juraska M, Huang Y, Zhuang Y, Fong Y, Carpp LN, Self SG, Chambonneau L, Small R, Jackson N, Noriega F, Gilbert PB. Neutralizing Antibody Correlates Analysis of Tetravalent Dengue Vaccine Efficacy Trials in Asia and Latin America. J Infect Dis. 2018 Feb 14;217(5):742-753. doi: 10.1093/infdis/jix609. PMID 29194547
- [Background] Arredondo-Garcia JL, Hadinegoro SR, Reynales H, Chua MN, Rivera Medina DM, Chotpitayasunondh T, Tran NH, Deseda CC, Wirawan DN, Cortes Supelano M, Frago C, Langevin E, Coronel D, Laot T, Perroud AP, Sanchez L, Bonaparte M, Limkittikul K, Chansinghakul D, Gailhardou S, Noriega F, Wartel TA, Bouckenooghe A, Zambrano B; CYD-TDV Dengue Vaccine Study Group. Four-year safety follow-up of the tetravalent dengue vaccine efficacy randomized controlled trials in Asia and Latin America. Clin Microbiol Infect. 2018 Jul;24(7):755-763. doi: 10.1016/j.cmi.2018.01.018. Epub 2018 Feb 8. PMID 29408333
- [Background] Thomas SJ, Yoon IK. A review of Dengvaxia(R): development to deployment. Hum Vaccin Immunother. 2019;15(10):2295-2314. doi: 10.1080/21645515.2019.1658503. Epub 2019 Oct 7. PMID 31589551
- [Background] Friberg H, Beaumier CM, Park S, Pazoles P, Endy TP, Mathew A, Currier JR, Jarman RG, Anderson KB, Hatch S, Thomas SJ, Rothman AL. Protective versus pathologic pre-exposure cytokine profiles in dengue virus infection. PLoS Negl Trop Dis. 2018 Dec 17;12(12):e0006975. doi: 10.1371/journal.pntd.0006975. eCollection 2018 Dec. PMID 30557313
- [Background] Rothman AL. Cellular immunology of sequential dengue virus infection and its role in disease pathogenesis. Curr Top Microbiol Immunol. 2010;338:83-98. doi: 10.1007/978-3-642-02215-9_7. PMID 19802580
- [Background] Ng KH, Zhang SL, Tan HC, Kwek SS, Sessions OM, Chan CY, Liu ID, Lee CK, Tambyah PA, Ooi EE, Yap HK. Persistent Dengue Infection in an Immunosuppressed Patient Reveals the Roles of Humoral and Cellular Immune Responses in Virus Clearance. Cell Host Microbe. 2019 Nov 13;26(5):601-605.e3. doi: 10.1016/j.chom.2019.10.005. Epub 2019 Oct 29. PMID 31676304
- [Background] Ong EZ, Gan ES, de Alwis R, Wijaya L, Ong XM, Zhang M, Wong AW, Cheung YB, Zellweger RM, Ooi EE, Low JG. Genomic signature of early T-cell response is associated with lower antibody titer threshold for sterilizing immunity. Antiviral Res. 2019 Jun;166:35-41. doi: 10.1016/j.antiviral.2019.03.013. Epub 2019 Mar 30. PMID 30940521
- [Background] Barrett ADT. The reemergence of yellow fever. Science. 2018 Aug 31;361(6405):847-848. doi: 10.1126/science.aau8225. Epub 2018 Aug 23. No abstract available. PMID 30139914
- [Background] Akondy RS, Monson ND, Miller JD, Edupuganti S, Teuwen D, Wu H, Quyyumi F, Garg S, Altman JD, Del Rio C, Keyserling HL, Ploss A, Rice CM, Orenstein WA, Mulligan MJ, Ahmed R. The yellow fever virus vaccine induces a broad and polyfunctional human memory CD8+ T cell response. J Immunol. 2009 Dec 15;183(12):7919-30. doi: 10.4049/jimmunol.0803903. PMID 19933869
- [Background] Gaucher D, Therrien R, Kettaf N, Angermann BR, Boucher G, Filali-Mouhim A, Moser JM, Mehta RS, Drake DR 3rd, Castro E, Akondy R, Rinfret A, Yassine-Diab B, Said EA, Chouikh Y, Cameron MJ, Clum R, Kelvin D, Somogyi R, Greller LD, Balderas RS, Wilkinson P, Pantaleo G, Tartaglia J, Haddad EK, Sekaly RP. Yellow fever vaccine induces integrated multilineage and polyfunctional immune responses. J Exp Med. 2008 Dec 22;205(13):3119-31. doi: 10.1084/jem.20082292. Epub 2008 Dec 1. PMID 19047440
- [Background] Querec TD, Akondy RS, Lee EK, Cao W, Nakaya HI, Teuwen D, Pirani A, Gernert K, Deng J, Marzolf B, Kennedy K, Wu H, Bennouna S, Oluoch H, Miller J, Vencio RZ, Mulligan M, Aderem A, Ahmed R, Pulendran B. Systems biology approach predicts immunogenicity of the yellow fever vaccine in humans. Nat Immunol. 2009 Jan;10(1):116-125. doi: 10.1038/ni.1688. Epub 2008 Nov 23. PMID 19029902
- [Background] Pulendran B. Learning immunology from the yellow fever vaccine: innate immunity to systems vaccinology. Nat Rev Immunol. 2009 Oct;9(10):741-7. doi: 10.1038/nri2629. Epub 2009 Sep 18. PMID 19763148
- [Background] Li X, Ma SJ, Liu X, Jiang LN, Zhou JH, Xiong YQ, Ding H, Chen Q. Immunogenicity and safety of currently available Japanese encephalitis vaccines: a systematic review. Hum Vaccin Immunother. 2014;10(12):3579-93. doi: 10.4161/21645515.2014.980197. PMID 25668666
- [Background] Monath TP, Seligman SJ, Robertson JS, Guy B, Hayes EB, Condit RC, Excler JL, Mac LM, Carbery B, Chen RT; Brighton Collaboration Viral Vector Vaccines Safety Working Group (V3SWG). Live virus vaccines based on a yellow fever vaccine backbone: standardized template with key considerations for a risk/benefit assessment. Vaccine. 2015 Jan 1;33(1):62-72. doi: 10.1016/j.vaccine.2014.10.004. Epub 2014 Oct 27. PMID 25446819
- [Background] Mishra N, Boudewijns R, Schmid MA, Marques RE, Sharma S, Neyts J, Dallmeier K. A Chimeric Japanese Encephalitis Vaccine Protects against Lethal Yellow Fever Virus Infection without Inducing Neutralizing Antibodies. mBio. 2020 Apr 7;11(2):e02494-19. doi: 10.1128/mBio.02494-19. PMID 32265332
- [Background] Nasveld PE, Marjason J, Bennett S, Aaskov J, Elliott S, McCarthy K, Kanesa-Thasan N, Feroldi E, Reid M. Concomitant or sequential administration of live attenuated Japanese encephalitis chimeric virus vaccine and yellow fever 17D vaccine: randomized double-blind phase II evaluation of safety and immunogenicity. Hum Vaccin. 2010 Nov;6(11):906-14. doi: 10.4161/hv.6.11.12854. Epub 2010 Nov 1. PMID 20864814
- [Background] Singh R, Rothman AL, Potts J, Guirakhoo F, Ennis FA, Green S. Sequential immunization with heterologous chimeric flaviviruses induces broad-spectrum cross-reactive CD8+ T cell responses. J Infect Dis. 2010 Jul 15;202(2):223-33. doi: 10.1086/653486. PMID 20536361
- [Background] Low JG, Ng JHJ, Ong EZ, Kalimuddin S, Wijaya L, Chan YFZ, Ng DHL, Tan HC, Baglody A, Chionh YH, Lee DCP, Budigi Y, Sasisekharan R, Ooi EE. Phase 1 Trial of a Therapeutic Anti-Yellow Fever Virus Human Antibody. N Engl J Med. 2020 Jul 30;383(5):452-459. doi: 10.1056/NEJMoa2000226. PMID 32726531
- [Background] Chan KR, Wang X, Saron WAA, Gan ES, Tan HC, Mok DZL, Zhang SL, Lee YH, Liang C, Wijaya L, Ghosh S, Cheung YB, Tannenbaum SR, Abraham SN, St John AL, Low JGH, Ooi EE. Cross-reactive antibodies enhance live attenuated virus infection for increased immunogenicity. Nat Microbiol. 2016 Sep 19;1(12):16164. doi: 10.1038/nmicrobiol.2016.164. PMID 27642668
- [Background] Monath TP, Guirakhoo F, Nichols R, Yoksan S, Schrader R, Murphy C, Blum P, Woodward S, McCarthy K, Mathis D, Johnson C, Bedford P. Chimeric live, attenuated vaccine against Japanese encephalitis (ChimeriVax-JE): phase 2 clinical trials for safety and immunogenicity, effect of vaccine dose and schedule, and memory response to challenge with inactivated Japanese encephalitis antigen. J Infect Dis. 2003 Oct 15;188(8):1213-30. doi: 10.1086/378356. Epub 2003 Oct 3. PMID 14551893
- [Derived] Kalimuddin S, Tham CYL, Chan YFZ, Hang SK, Kunasegaran K, Chia A, Chan CYY, Ng DHL, Sim JXY, Tan HC, Syenina A, Ngoh AQ, Hamis NZ, Chew V, Leong YS, Yee JX, Low JG, Chan KR, Ong EZ, Bertoletti A, Ooi EE. Vaccine-induced T cell responses control Orthoflavivirus challenge infection without neutralizing antibodies in humans. Nat Microbiol. 2025 Feb;10(2):374-387. doi: 10.1038/s41564-024-01903-7. Epub 2025 Jan 10. PMID 39794472
- [Derived] Kalimuddin S, Chan YFZ, Sessions OM, Chan KR, Ong EZ, Low JG, Bertoletti A, Ooi EE. An experimental medicine decipher of a minimum correlate of cellular immunity: Study protocol for a double-blind randomized controlled trial. Front Immunol. 2023 Mar 10;14:1135979. doi: 10.3389/fimmu.2023.1135979. eCollection 2023. PMID 36969244
- See also: Centers for Disease Control and Prevention. Yellow Fever 2018 — http://wwwnc.cdc.gov/travel/yellowbook/2018/infectious-diseases-related-to-travel/yellow-fever.